CLINICAL TRIAL: NCT00890643
Title: Effect of Prazosin on Neurophysiologic Responses and Cognitive Performance in PTSD
Brief Title: Effect of Prazosin on Neurophysiology and Cognition in Post-Traumatic Stress Disorder (PTSD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary investigator left VA employment
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MHBA-018-08S
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Stress disorders, post-traumatic; Combat Disorders; prazosin; cognition; neurophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Prazosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Persons with PTSD
  Interventions: Drug: prazosin hydrochloride
- Arm 2 (Placebo Comparator): Persons with PTSD
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: prazosin hydrochloride — prazosin 1-20 mg/day in divided doses
  Other Names: Minipress
  Arms: Arm 1
Drug: placebo — placebo
  Arms: Arm 2

SUMMARY:
In this study, the investigators are looking at how PTSD affects things such as memory, attention, reaction to sounds, eye movements, and heart rate. The investigators are also studying whether a medication called prazosin has an effect on these things.

DETAILED DESCRIPTION:
Converging lines of evidence suggest that central nor adrenergic function is perturbed in PTSD. Placebo-controlled trials demonstrate that the centrally acting alpha-1 antagonist prazosin is clinically effective for several core symptoms of PTSD in combat veterans. However, no detailed assessment of the impact of prazosin on human neurophysiology and cognition have been conducted. Our hypotheses are based on studies that demonstrate (1) the importance of central adrenergic receptors in regulating fundamental neurophysiologic and cognitive functions, (2) the alteration of these functions in PTSD, and (3) the efficacy of prazosin in improving the clinical symptoms of PTSD. The primary objective of this study is to measure the subtle neurocognitive and neurophysiologic effects on prazosin in combat veterans with PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Exposure to one or more life-threatening war zone trauma events;
* DSM-IV diagnosis of PTSD derived from the Clinician-Administered PTSD Scale (CAPS), CAPS total score greater than or equal to 50;
* CAPS recurrent distressing dreams item score greater than or equal to 5 (of a maximum score of 8), with a frequency rating greater than or equal to 2 (of 4);
* stable dose of non-exclusionary medications and psychotherapeutic treatment for at least 4 weeks prior to randomization;
* good general medical health;
* female participants must agree to use a reliable form of birth control throughout study.

Exclusion Criteria:

* Acute or unstable chronic medical illness;
* diagnosis of current schizophrenia, schizoaffective disorder, psychotic disorder not otherwise specified, bipolar disorder, delirium, or cognitive disorder;
* severe psychiatric instability or severe situational life crises;
* substance dependence disorder currently or in past 3 months;
* current cocaine or stimulant abuse or evidence of acute intoxication on alcohol or nonprescribed medication;
* allergy or previous adverse reaction to prazosin or other alpha-1 adrenergic antagonists;
* serious head injury with loss of consciousness of greater than 30 minutes;
* current diagnosis of seizure disorder;
* current use of prazosin or other alpha-1 adrenergic antagonists;
* current use of atypical antipsychotic medication;
* stimulants or alternative medications with stimulant properties (e.g. ephedra), certain exposure therapies must be completed at least 4 weeks before baseline;
* certain medications (trazodone, erectile disfunction medications) are not allowed or are restricted during the study;
* women must not be pregnant or nursing during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Responses to acoustic startle and prepulse inhibition of acoustic startle | baseline, week 2, week 8

SECONDARY OUTCOMES:
Heart rate variability | baseline, week 2, week 8
Pennsylvania Computerized Neurocognitive Battery (CNB) | baseline, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Dorcas J. Dobie, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States